CLINICAL TRIAL: NCT06833060
Title: Exploratory Clinical Study of a Laser-OCT Integrated System With Eye Tracking to Treat Glaucoma and OHT With Transscleral Selective Laser Trabeculoplasty Technology A Pilot Study
Brief Title: Transscleral Selective Laser Trabeculoplasty Project
Acronym: TSLT project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lumibird Medical (Quantel Medical, Ellex Medical, Optotek) (Industry)
Collaborators: Quantel Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TSLT-001-2023
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma,Open-Angle; Ocular Hypertension (OH)
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transscleral Selective Laser trabeculoplasty treatment (Experimental): The Glaucoma or Ocular Hypertension participants will be treated using Transscleral Selective Trabeculoplasty laser device.
  Interventions: Device: Selective Laser Trabeculoplasty

INTERVENTIONS:
Device: Selective Laser Trabeculoplasty — Treatment of Glaucoma or Ocular Hypertension participants using Transscleral Selective Laser Trabeculoplasty
  Other Names: Transscleral Selective Laser Trabeculoplasty

SUMMARY:
The purpose of this clinical trial is to determine how safe and effective (how well it works) the ELLEX TSLT device is for the treatment of Glaucoma and Ocular Hypertension using Transscleral Selective Laser Trabeculoplasty.

Selective Laser Trabeculoplasty (SLT) is a type of laser therapy that uses short pulses of low-energy light to lower eye pressure. This treatment uses a lens in contact with the front part of the eye (called cornea) which may lead to complications. Transscleral Selective Laser Trabeculoplasty allows the doctor to perform the laser treatment without the lens coming into contact with the cornea, potentially offering a simpler, quicker and safer approach for both participants and doctors.

Participants will be required to attend four study visits. The first visit will assess the disease, the second will involve the TSLT laser treatment for the participant's condition (glaucoma or ocular hypertension), and the final two visits, at 1 day and 30 days post-treatment, will evaluate the treatment's efficacy and the procedure's safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older with OAG or OHT who are clinical candidates for routine SLT.
* Mild to moderate OAG (defined as a mean deviation on the Humhprey Field Analyzer [HFA] > -12.0 dB), resulting from primary open-angle glaucoma (POAG), or pseudoexfoliative glaucoma
* OHT with open angles warranting IOP-lowering treatment
* IOP ≥ 22mmHg or ≤ 35mmHg (after washout of any IOP-lowering medications)
* Gonioscopically visible scleral spur for 360 degrees without indentation
* Ability to visualize the peri-limbal sclera for 360 degrees (using a manual elevation of the lid)
* Willing and able to participate in the 60 days +/-5 days study, to comply with the study procedures and to adhere to the follow-up schedule.
* Participant capable of giving informed consent

Exclusion Criteria:

* Contraindications to conventional SLT (e.g. corneal abnormalities etc.)
* Angle Closure Glaucoma
* Congenital or developmental glaucoma
* Secondary glaucoma included pigmentary glaucoma
* Inability to conduct a reliable visual field (defined as fixation losses, false positives or false negatives greater than 33%)
* Presence of any peripheral anterior synechiae (PAS) in the study eye
* Any of the following visual field findings using the Humphrey visual field analyzer:

  * A HFA MD of worse than -12dB
  * Greater than or equal to 75% of points depressed below the 5% level and greater than or equal to 50% of points depressed below the 1% level on the PD plot
  * At least 50% of points (i.e., 2 or more) within the central 5 degrees with a sensitivity ≤0dB on the decibel plot
  * Points within the central 5 degrees of fixation with a sensitivity <15 dB in both hemifields on the decibel plot
  * A visual field MD of worse than -12dB in the fellow eye
* Cup: Disc Ratio more than 0.8
* More than two hypotensive medications required (combination drops are considered 2 medications)
* Prior incisional or laser glaucoma surgery (including previous SLT) in the study eye
* Prior corneal refractive surgery
* Complicated cataract surgery ≤ 6 months prior to enrollment
* Presence of visually significant cataract in the opinion of the investigator
* Clinically significant disease in either eye as determined by the Investigator
* Clinically significant amblyopia in either eye
* Dense pigmentation or hemorrhage in the peri-limbal conjunctiva or anterior sclera, Pigmented Pinguecula and Pterigium
* Women who are pregnant or may become pregnant during the course of the study
* In the opinion of the investigator the participant might require other ocular surgery within the 12-months, unless for further reduction of their IOP.
* Concurrent treatment with topical, nasal, inhaled or systemic steroids.
* Uncontrolled systemic disease that could impact the ability of the participant to attend follow up visits as per the discretion of the investigator
* Participation in another clinical study
* Protected or vulnerable subjects (including but not limited to people with impaired intellectual functioning or mental illness, prisoners, terminally ill subjects, immunocompromised…)
* People not able to read and understand the informed consent
* People not able to read and understand English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Treatment-Related Adverse Events | From treatment to 30 days after
Intensity of Treatment-Related Adverse Events | From treatment to 30 days after

SECONDARY OUTCOMES:
Ability of the TSLT device to decrease the patient's Intraocular pressure | 30 days after treatment
  IOP reduction after TSLT treatment will be compared to the 20% threshold efficacy point as defined in the SLT literature
Benchmark with the available Direct Selective Laser Trabecuplasty studies data | 30 days after treatment
Trabecular meshwork targeting | Day of treatment
  Demonstration of the right targeting of the trabecular meshwork by the device using OCT images.
Usability assessment | Day of treatment
  Evaluation of how easily users can interact with the device and how this device can improve the treatment delivery (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. CASSON, MBBS (Hons), M.Biostat, DPhil, Principal Investigator — Royal Adelaide Hospital - Harley Eye Clinic; Mario de La TORRE, Prof. Dr. med., Study Director — Lumibird Medical (Quantel Medical, Ellex Medical, Optotek)
Locations (1):
- Central Adelaide Local Health Network - Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No